CLINICAL TRIAL: NCT05178732
Title: The Effect of Menstrual Cycle Phase and Protein Dose on Muscle Protein Synthesis in Response to Exercise in Young Females
Brief Title: The Effect of Menstrual Cycle Phase and Protein Dose on Muscle Protein Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: P.volve (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 21-10-20-B-03
Record Dates: First submitted 2021-12-07; First posted 2022-01-05 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Muscle Protein Synthesis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Protein dose 1 and early (Experimental)
  Interventions: Dietary Supplement: Dose of protein; Other: Menstrual cycle phase
- Protein dose 1 and late (Experimental)
  Interventions: Dietary Supplement: Dose of protein; Other: Menstrual cycle phase
- Protein dose 2 and early (Experimental)
  Interventions: Dietary Supplement: Dose of protein; Other: Menstrual cycle phase
- Protein dose 2 and late (Experimental)
  Interventions: Dietary Supplement: Dose of protein; Other: Menstrual cycle phase
- Protein dose 3 and early (Experimental)
  Interventions: Dietary Supplement: Dose of protein; Other: Menstrual cycle phase
- Protein dose 3 and late (Experimental)
  Interventions: Dietary Supplement: Dose of protein; Other: Menstrual cycle phase

INTERVENTIONS:
Dietary Supplement: Dose of protein — One of three protein doses provided
Other: Menstrual cycle phase — Different phase of the menstrual cycle

SUMMARY:
Adaptation to resistance exercise requires maximal rates of muscle protein synthesis, which can be achieved with post-exercise ingestion of ~20g of protein. These recommendations are based on studies in males and responses in females may vary.

Muscle recovery is related to the ability to build new muscle protein from amino acids (muscle protein synthesis). This response is thought to be impacted in females by hormones that fluctuate across different phases of the menstrual cycle. However, the effect of menstrual cycle phase on muscle protein synthesis is not known.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 30
* Recreationally active
* Regular menstrual cycle

Exclusion Criteria:

* Smoking
* Metabolic disease
* Any motor disorder
* Use of over-the-counter pharmaceuticals, during the study.
* Pomegranate, milk or lidocaine allergy
* Taken contraceptives in the past 3 months
* Irregular menstrual cycle (less than 9 cycles per year and a length not between 21-35 days)
* Post-menopausal women
* Pregnancy and lactation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-16 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis | 7.5 hours
  The rate of synthesis of new muscle protein

SECONDARY OUTCOMES:
Plasma amino acid kinetics | 7.5 hours
  The appearance of amino acids in the circulation.
Serum insulin concentrations | 7.5 hours
  Basal and postprandial concentrations of serum insulin
Blood flow | 7.5 hours
  Basal and postprandial blood flow using ultrasound
Sex hormone concentrations | 5 minutes
  Serum oestrogen and progesterone
Gene expression | 7.5 hours
  Gene expression of muscle samples using RNA extraction
Blood glucose | 7.5 hours
  Basal and postprandial concentrations of blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: Francis Stephens, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No